CLINICAL TRIAL: NCT03374657
Title: An Open-label First-in-human Single Ascending Dose Study to Explore Safety, Tolerability and Efficacy of Subretinal Administration of CPK850 Gene Therapy in Patients With Retinitis Pigmentosa Due to Mutations in the Retinaldehyde Binding Protein 1 (RLBP1) Gene
Brief Title: A First-in-human, Proof of Concept Study of CPK850 in Patients With RLBP1 Retinitis Pigmentosa
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CCPK850X2202; 2016-002696-10 (EudraCT Number)
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Retinitis Pigmentosa
Keywords: Clinical trials, dark adaptation, gene therapy, RLBP1 mutation, retinitis pigmentosa.
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: This is a non-confirmatory, open-label single ascending dose gene replacement-therapy study to assess safety, tolerability and efficacy of CPK850 in patients with RLBP1 retinitis pigmentosa due to biallelic mutations in the RLBP1 gene. The trial design uses a staggered patient enrollment.
Who Masked: Outcomes Assessor
Masking Description: This is a partially masked study. The patients will not be masked. The treating physicians and personnel at the surgical location (surgeons, anesthesiologist, operating room personnel and others) will not be masked.
  At the clinical sites, there will be an unmasked ophthalmologist. The remaining assessors at the clinical sites (ophthalmologist, study nurse, ophthalmic technician, etc) doing the ophthalmic examinations should be masked to the study (treated) eye.
  The following unmasked sponsor roles are required for this study:
  Sponsor clinical staff required to assist in the management and re-supply of investigational drug product.
  The independent committee assessing unmasked interim results and the independent analysis team.
  All other sponsor staff will stay masked to treatment assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CPK Dose 1 (lowest dose) (Experimental): CPK850, one subretinal injection to the study eye
  Interventions: Biological: CPK850
- CPK Dose 2 (next lowest dose) (Experimental): CPK850, one subretinal injection to the study eye
  Interventions: Biological: CPK850
- CPK Dose 3 (third lowest dose) (Experimental): CPK850, one subretinal injection to the study eye
  Interventions: Biological: CPK850
- CPK Dose 4 (highest dose) (Experimental): CPK850, one subretinal injection to the study eye
  Interventions: Biological: CPK850

INTERVENTIONS:
Biological: CPK850 — In one of 4 dose levels administered via subretinal injection under anesthesia

SUMMARY:
The purpose of this first-in-human study is to explore the maximum tolerated dose (MTD) of CPK850 as determined by the single ascending dose ranging portion of the study. This study will also evaluate the safety and potential efficacy of CPK850 on improving visual function in patients with decreased visual function from RLBP1 retinitis pigmentosa due to biallelic mutations in the RLBP1 gene.

DETAILED DESCRIPTION:
This study will potentially include 4 cohorts with a minimum of 3 patients per cohort. This trial design used a staggered patient enrollment with continuous data reviews to limit as much unforeseen risk as possible prior to enrolling each patient in each cohort or initiating another cohort. Only one eye (designated as the study or treated eye) will be dosed per patient. Each patient will be followed for 5 years after the subretinal injection of CPK850.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 70 years inclusive.
* The visual acuity in the study eye at the screening 1 visit should be no better than 60 ETDRS letters.
* Clinical diagnosis of Bothnia dystrophy, Newfoundland rod-cone dystrophy or other progressive retinitis pigmentosa phenotype with mutations in the RLBP1 gene verified by genetic testing.
* Visible photoreceptor (outer nuclear) and Retinal Pigment Epithelium (RPE) layers on standard OCT scan in the study eye at the screening 1 visit.

Exclusion Criteria:

* History of hypersensitivity to the study drug or to drugs of similar classes or to any of the medications required in the perioperative period.
* Pre-existing eye conditions that would preclude the planned surgery or interfere with the interpretation of study endpoints
* Any contraindication to the planned surgery or anesthesia as determined by the treating physician (surgeon, anesthesiologist, internist, or designee).
* Women who are pregnant, or lactating or women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for two months after treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs) and deaths | Up to year 5
  Safety events
Number of responders in dark adaptation | Screening/baseline up to year 1
  A patient is considered a responder if sensitivity recovery values at 1 hour post-bleach are observed to be outside of the patient's prediction interval at ≥2 consecutive post-treatment visits within one year after treatment.

SECONDARY OUTCOMES:
Number of patients with recovery of the cone system | Screening/baseline up to year 1
  cone recovery during dark adaptation
Number of patients with improvement in rod function in the treated eye vs the untreated eye | Screening/baseline up to year 1
  rod function during dark adaptation
Change from screening/baseline in Visual field perimetry mean deviation | Screening/baseline up to year 1
  Assessed using automated static perimetry
Change from screening/baseline in Total contrast sensitivity score | Screening/baseline up to year 1
  Contrast sensitivity (ie, the ability to detect relatively dim objects) will be assessed
Change from screening/baseline in Light-adapted microperimetry sensitivity | Screening/baseline up to year 1
  Assessed using standard microperimetry equipment
Change from screening/baseline in the local electrical activity of the retina | Screening/baseline up to year 1
  Assessed using a system designed to record multifocal electroretinogram (ERG) responses from a number of locations at one time
Change from screening/baseline in the electrical activity of the retina | Screening/baseline up to year 1
  Assessed using a system designed to record full-field electroretinogram (ERG) responses with Ganzfeld stimulation.
Change from screening/baseline in Reading speed | Screening/baseline up to year 1
  Assessed using standard reading speed charts
Change from screening/baseline in eye dominance | Screening/baseline up to year 1
  Dominant eye for viewing targets at distance
Change from screening/baseline in Change from baseline in mobility test scores | Screening/baseline up to year 1
  Assessed using a system designed to measure the ability to navigate obstacles in a maze-like environment under varying light conditions
Change from screening/baseline in the National Eye Institute - Visual function questionnaire 25 (NEI-VFQ 25) composite score | Screening/baseline up to year 1
  Questionnaire completed by the participant to measure the influence of visual impairment on quality of life
Change from screening/baseline in the low luminance questionnaire (LLQ) responses | Screening/baseline up to year 1
  Questionnaire completed by the participant to assess visual problems under low luminance conditions, including nighttime

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Kvanta A, Rangaswamy N, Holopigian K, Watters C, Jennings N, Liew MSH, Bigelow C, Grosskreutz C, Burstedt M, Venkataraman A, Westman S, Geirsdottir A, Stasi K, Andre H. Interim safety and efficacy of gene therapy for RLBP1-associated retinal dystrophy: a phase 1/2 trial. Nat Commun. 2024 Sep 10;15(1):7438. doi: 10.1038/s41467-024-51575-4. PMID 39256350